CLINICAL TRIAL: NCT02005497
Title: Increasing Implementation of Evidence-based Interventions at Low-wage Worksites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Peggy Hannon, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 45447-EJ; 1R01CA160217 (NIH)
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Cancer; Health Promotion
Keywords: Cancer prevention and control; Health promotion; Workplace; Dissemination; Implementation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HealthLinks (Experimental): Worksites in this arm will receive the standard HealthLinks intervention protocol, which includes on-site consulting, toolkits, and support via telephone and email to implement a worksite wellness program and adopt evidence-based practices.
  Interventions: Other: HealthLinks
- HealthLinks+ (Active Comparator): Worksites in this arm will receive the standard HealthLinks intervention protocol, which includes on-site consulting, toolkits, and support via telephone and email plus support to form a worker wellness committee to implement a worksite wellness program and adopt evidence-based practices.
  Interventions: Other: HealthLinks
- Delayed Control (No Intervention): Worksites in this arm will not receive an intervention during the study. After they have provided their final follow-up data, they will receive the HealthLinks intervention.

INTERVENTIONS:
Other: HealthLinks
  Arms: HealthLinks; HealthLinks+

SUMMARY:
The proposed project will answer key questions about implementing evidence-based health promotion interventions at small and low-wage worksites. Small, low-wage worksites will be randomized to receive HealthLinks (a free American Cancer Society program to disseminate evidence-based interventions), HealthLinks+ (which will include creating worksite wellness committees as part of the program), or to serve in a delayed control group. This approach will identify successful strategies for implementing evidence-based interventions at low-wage worksites to improve workers' cancer screening, healthy eating, physical activity, and tobacco cessation.

DETAILED DESCRIPTION:
Cancer and other chronic diseases are leading killers and disablers in the United States, and low-income Americans are at high risk for these diseases. Multiple evidence-based interventions (EBIs) exist to improve chronic disease risk behaviors, such as cancer screening, healthy eating, physical activity, and tobacco cessation, yet EBI reach to community settings is poor. Among community settings for reaching low-income adults, worksites stand out because most low-income adults are employed, but worksite implementation of health-promoting EBIs is low. Half of American workers work in small or low-wage worksites, where implementation of these EBIs and readiness to implement are especially low. Even though decision-makers at these worksites are often motivated to promote worker health, they usually have no dedicated wellness staff and face three major barriers in implementing EBIs: 1) lack of awareness of the potential benefits of EBIs, 2) lack of knowledge to choose EBIs, and 3) lack of financial and personnel resources to implement EBIs. Non-profit organizations and others who would assist these worksites face their own barriers. Organizational readiness to implement EBIs is not well understood, and few validated measures are available, especially for worksites. Without reliable and valid measures of worksite readiness, those who would assist them have difficulty: a) identifying worksites that are ready, and b) helping decision-makers get ready to increase their odds of implementation success. The proposed research will address both sets of barriers and contribute to dissemination and implementation research by testing the efficacy of a worksite EBI dissemination program, HealthLinks, developed in partnership with the American Cancer Society, a non-profit organization operating nationwide. HealthLinks is based on Greenhalgh's diffusion of innovations framework and Rogers' diffusion of innovations theory and addresses small and low-wage worksites' barriers by providing free on-site information and recommendations for EBIs and by providing free on-site programs and temporary staffing to assist implementation. We will test HealthLinks via a 3-arm randomized controlled trial. Worksites will receive either 1) HealthLinks, or 2) an enhanced version of HealthLinks that addresses small worksites' lack of personnel by adding worker wellness committees, or will 3) serve in a delayed control group that receives HealthLinks at study end. We will measure worksites' EBI implementation at baseline, 12 months (at the end of the intervention period), and 24 months (to assess maintenance one year after the intervention ends). This design will test the effectiveness of both HealthLinks and of worker wellness committees. We will also measure the effect of both on workers' health behaviors at baseline, 12 months, and 24 months. Finally, we will develop, pilot-test, and validate a measure of worksite readiness to implement EBIs.

ELIGIBILITY:
Inclusion Criteria (for worksites):

* 20-200 employees
* In one of the following industries: accommodation and food services; arts, entertainment, and recreation; educational services, health care and social assistance, other services excluding public administration, retail trade
* Located in King County, Washington State

Exclusion Criteria:

* Has a wellness committee
* Fewer than 20% of workers report to a physical worksite

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-12; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Worksite implementation of evidence-based health promotion interventions | up to 24 months
  The intervention being tested promotes a package of evidence-based health promotion interventions. The primary outcome is the proportion of these interventions the worksites are implementing at each time-point assessed.

SECONDARY OUTCOMES:
Workers' health behaviors related to cancer screening, nutrition, physical activity, and tobacco use | Measured at baseline, 12 months, and 24 months
  Workers at participating worksites will complete brief surveys at each time-point assessed that measure their health behaviors related to breast, cervical, and colon cancer screening, healthy eating, physical activity, and tobacco use/cessation.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret A Hannon, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Health Promotion Research Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hannon PA, Harris JR, Sopher CJ, Kuniyuki A, Ghosh DL, Henderson S, Martin DP, Weaver MR, Williams B, Albano DL, Meischke H, Diehr P, Lichiello P, Hammerback KE, Parks MR, Forehand M. Improving low-wage, midsized employers' health promotion practices: a randomized controlled trial. Am J Prev Med. 2012 Aug;43(2):125-33. doi: 10.1016/j.amepre.2012.04.014. PMID 22813676
- [Background] Laing SS, Hannon PA, Talburt A, Kimpe S, Williams B, Harris JR. Increasing evidence-based workplace health promotion best practices in small and low-wage companies, Mason County, Washington, 2009. Prev Chronic Dis. 2012;9:E83. Epub 2012 Apr 5. PMID 22480612
- [Background] Hannon PA, Hammerback K, Allen CL, Parrish AT, Chan KG, Kohn MJ, Teague S, Beresford SA, Helfrich CD, Harris JR. HealthLinks randomized controlled trial: Design and baseline results. Contemp Clin Trials. 2016 May;48:1-11. doi: 10.1016/j.cct.2016.02.011. Epub 2016 Mar 2. PMID 26946121
- [Background] Hannon PA, Helfrich CD, Chan KG, Allen CL, Hammerback K, Kohn MJ, Parrish AT, Weiner BJ, Harris JR. Development and Pilot Test of the Workplace Readiness Questionnaire, a Theory-Based Instrument to Measure Small Workplaces' Readiness to Implement Wellness Programs. Am J Health Promot. 2017 Jan;31(1):67-75. doi: 10.4278/ajhp.141204-QUAN-604. Epub 2016 Nov 17. PMID 26389975
- [Background] Hammerback K, Hannon PA, Harris JR, Clegg-Thorp C, Kohn M, Parrish A. Perspectives on Workplace Health Promotion Among Employees in Low-Wage Industries. Am J Health Promot. 2015 Jul-Aug;29(6):384-92. doi: 10.4278/ajhp.130924-QUAL-495. Epub 2014 Aug 27. PMID 25162321
- [Derived] Harris JR, Kava CM, Chan KCG, Kohn MJ, Hammerback K, Parrish AT, Helfrich CD, Hannon PA. Pathways to Employee Outcomes in a Workplace Health Promotion Program. Am J Health Promot. 2022 May;36(4):662-672. doi: 10.1177/08901171211066898. Epub 2022 Jan 4. PMID 34983199